CLINICAL TRIAL: NCT03020901
Title: 100000cases Real World Research of the Safety, Efficacy Reassessment, and Bacterial Resistance Monitoring of Teicoplanin for Injection After Listing
Brief Title: the Clinical Trial of Teicoplanin for Injection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: FM-P5-2016052501
Record Dates: First submitted 2017-01-06; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases | interventions — Teicoplanin; Injections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Teicoplanin for Injection — Use Teicoplanin for Injection
  Other Names: Ta Ge Shi

SUMMARY:
1. Primary study endpoint Security Effectiveness
2. Secondary study endpoint Extensive use of population characteristics Clinical drug characteristics appropriate crowd characteristics Adverse reactions susceptible population characteristics Reveal rare, new, unanticipated and long-term adverse drug reactions bacterial resistance Explore the advantages of teicoplanin in combination with other antimicrobial agents Explore the opportunistic use of teicoplanin for injection

DETAILED DESCRIPTION:
Research purposes

1. To explore the safety and efficacy of different doses of teicoplanin for injection in the real world
2. To explore the characteristics of different doses of teicoplanin for injection, the clinical characteristics of drug use and repeated use of bacterial resistance;
3. Reveal rare or even very rare, new, unanticipated, and adverse drug reactions associated with long-term use;
4. To explore the advantages of different doses of teicoplanin in combination with other antimicrobial agents;
5. To explore the use of teicoplanin in the treatment of infectious diseases on the rational use of drugs time;
6. To reveal the risk factors of adverse reactions and susceptibility to people, to identify the characteristics of the crowd;
7. To investigate the clinical use of teicoplanin injection for the real situation, for further risk management, to expand the indications and expert consensus dose study to provide clinical clues and basis;
8. To provide reference for revision of clinical guidelines and consensus, clinical pathway design;
9. To further enhance the level of safe use of teicoplanin injection, basic medical support and market vitality.

Research design

1. National, large-scale, standardized, standardized, real-world research;
2. Prospective, single - arm open, non - interventional, registration, multi - center clinical study;
3. In the hospitals using teicoplanin for injection, 200 were selected on the basis of voluntary principles;
4. Registration of teicoplanin in patients with injection;
5. Target sample size of 100,000 cases;
6. Exemption from informed consent for ethical review applications;
7. Study of teicoplanin and large-scale data on the safety and effectiveness of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Prescription for teicoplanin in patients

Exclusion Criteria:

* NO

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prescription for teicoplanin in patients
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Bacterial clearance rate | 1-21 days after injection

IPD SHARING:
Plan to Share IPD: Undecided